CLINICAL TRIAL: NCT03930563
Title: Acute Beetroot Juice Supplementation and Peripheral Chemoreflex Sensitivity in Patients With Obstructive Sleep Apnea
Brief Title: Inorganic Nitrate and OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Darren P Casey, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 201812786
Record Dates: First submitted 2019-04-19; First posted 2019-04-29 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: inorganic nitrate; blood flow; Peripheral chemoreflex; Common carotid artery
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beetroot Juice Low (Experimental): Subjects will consume beetroot juice containing 250mg inorganic nitrate and 20mg nitrite dissolved in 120ml bottled water. Peripheral chemoreflex sensitivity as well as common carotid artery blood flow will be assessed before and after supplementation.
  Interventions: Dietary Supplement: Pre-beetroot juice supplementation; Dietary Supplement: Post-beetroot juice supplementation
- Beetroot Juice High (Experimental): Subjects will consume beetroot juice containing 500mg inorganic nitrate and 40mg nitrite dissolved in 120ml bottled water. Peripheral chemoreflex sensitivity as well as common carotid artery blood flow will be assessed before and after supplementation.
  Interventions: Dietary Supplement: Pre-beetroot juice supplementation; Dietary Supplement: Post-beetroot juice supplementation
- Beetroot Juice Placebo (Active Comparator): Subjects will consume beetroot juice devoid of inorganic nitrate and nitrite dissolved in 120ml bottled water. Peripheral chemoreflex sensitivity as well as common carotid artery blood flow will be assessed before and after supplementation.
  Interventions: Dietary Supplement: Pre-beetroot juice supplementation; Dietary Supplement: Post-beetroot juice supplementation

INTERVENTIONS:
Dietary Supplement: Pre-beetroot juice supplementation — Before administering beetroot juice to subjects.
Dietary Supplement: Post-beetroot juice supplementation — After administering beetroot juice to subjects.

SUMMARY:
The main purpose of this study is to determine if acute beetroot juice supplementation reduces peripheral chemoreflex sensitivity in patients with obstructive sleep apnea. All subjects will consume low-dose (BRL), higher-dose (BRH), and placebo (BRP) beetroot juice randomly on three independent study visits. Beetroot juice also improves blood flow thus, the investigators will also measure blood flow to the carotid chemoreceptors.

DETAILED DESCRIPTION:
Four-weeks of daily beetroot juice supplementation reduces peripheral chemoreflex sensitivity in healthy older adults who have 'normal' responses to acute hypoxia. Patients with obstructive sleep apnea have exaggerated peripheral chemoreflex sensitivity. It remains unknown if beetroot juice supplementation reduces peripheral chemoreflex sensitivity in patients with obstructive sleep apnea. Additionally, increasing blood flow to the peripheral chemoreceptors reduces sensitivity. Given that beetroot juice improves blood flow, the investigators will also measure common carotid artery blood flow at rest and during hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* OSA group: patients recently diagnosed with mild-to-moderate OSA
* Control group: healthy individuals

Exclusion Criteria:

* Diagnosis of heart disease
* Diagnosis of diabetes
* Diagnosis of any autonomic disorders
* Diagnosis of kidney disease
* Diagnosis of central sleep apnea
* Regular physical activity exceeding 30 minutes 3 days/week
* A body mass index ≥40 kg/m2
* Current or former use of a continuous positive airway pressure machine
* Current tobacco use
* Currently prescribed hormone replacement therapy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Changes in peripheral chemoreflex sensitivity | Before and after consuming all supplements (within three hours)
  The ventilatory response to acute hypoxia will be measured via pneumotachometer.

SECONDARY OUTCOMES:
Changes in common carotid artery blood flow | Before and after consuming all supplements (within three hours)
  Blood flow through the common carotid artery before and during hypoxia measured via Doppler ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Darren P Casey, PhD, Principal Investigator — University of Iowa
Locations (1):
- Medical Education Building, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No